CLINICAL TRIAL: NCT02756286
Title: Neurophysiological Attention Test (NAT) for Objective Assessment of Adult ADHD
Acronym: NAT-II
Status: Completed | Type: Observational
Sponsor: Think Now Incorporated (Industry)
Collaborators: University of California, Los Angeles (Other); University of California, Berkeley (Other); Oregon Health and Science University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gregory Simpson, Ph.D., Founder and Chief Scientific Officer, Think Now Incorporated
Other Study IDs: TNI-NAT-II; R44MH099709 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2016-04-29 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Electroencephalography; Attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHD: Adults with ADHD: NAT electroencephalography (EEG) test
  Interventions: Other: NAT electroencephalography (EEG) test
- Controls: Healthy adults without ADHD: NAT electroencephalography (EEG) test
  Interventions: Other: NAT electroencephalography (EEG) test

INTERVENTIONS:
Other: NAT electroencephalography (EEG) test — Individuals in both groups are asked to perform standard behavioral tests and an electroencephalography (EEG) test.

SUMMARY:
The purpose of this study is to refine a new assessment tool for Attention Deficit/Hyperactivity Disorder (ADHD) and then to test its validity (i.e. ability to discriminate between individuals with ADHD and healthy controls.

DETAILED DESCRIPTION:
The purpose of this study is to build upon the success the novel approach and software for analyzing electroencephalography (EEG) data to identify biomarkers of ADHD in adults by further refining the method. Then to test the ability of this new assessment tool to differentiate between adults with ADHD and healthy controls by comparing the classification accuracy of the metrics from the new tool to the classification accuracy of existing behavioral tests for ADHD.

ELIGIBILITY:
Inclusion Criteria:

Specific inclusion criteria for ADHD are:

1. meet established Diagnositic and Statistical Manual-5 criteria for ADHD predominately inattentive or combined subtype with clinically significant levels of impairment, diagnosed by structured clinical interview, the Mini International Neuropsychiatric Interview, and corroborating information
2. Clinical Global Impression-Severity (CGI-S) score ≥ 4 for ADHD
3. no lifetime history of DSM-5 bipolar disorder, psychotic disorder, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse, or substance dependence (except nicotine) as assessed with the Mini International Neuropsychiatric Interview (MINI).
4. able in the opinion of the investigator to complete all required study procedures.

Exclusion Criteria:

Exclusion criteria for both groups are:

1. History of diagnosis of childhood disorder other than ADHD (e.g. autism, dyslexia)
2. history of any general medical condition likely to require chronic use of medication with identified central nervous system (CNS) effects suspected to alter cognitive performance
3. history of seizure disorder, brain tumor, other major neurological disorder or head injury resulting in loss of consciousness
4. serious oxygen deprivation
5. current psychopathology requiring ongoing treatment with antipsychotic medications, mood stabilizers, benzodiazepines, or anticonvulsants
6. current untreated psychopathology which is rated to be primary in terms of severity (greater than ADHD severity)
7. current treatment with guanfacine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with Attention Deficit Hyperactivity Disorder (ADHD) from local clinics, clinicians, ADHD community resources in the area of each of the three participating Universities (UCLA, UCB, OHSU)
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
NAT Slow Fluctuation Test and Retest to assess change for Test Replicability | A single measurement is made for each individual at DAY 1 - the time of the brain wave (EEG) test; and a single measure is made again in each individual at least 30 days later (DAY 2) to identify any differences, to assess replicability of the measure.
  The NAT EEG test simultaneously generates 2 EEG values and 1 behavioral value that are used together as an assessment metric for ADHD. This is a one-time measure to assess its magnitude in ADHD vs Control.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory V Simpson, Ph.D., Principal Investigator — Think Now, Inc.
Locations (3):
- United States (3):
  - University of California Berkeley, Berkeley, California
  - UCLA Semel Institute, Los Angeles, California
  - Oregon Health & Science University, Portland, Oregon